CLINICAL TRIAL: NCT01188681
Title: A Phase 1b/2 Open Label Study to Evaluate the Safety and Efficacy of TRU-016 in Combination With Bendamustine vs. Bendamustine Alone in Patients With Relapsed Chronic Lymphocytic Leukemia
Brief Title: Safety and Efficacy Study of TRU-016 Plus Bendamustine vs. Bendamustine in Relapsed Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aptevo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16201
Record Dates: First submitted 2010-08-20; First posted 2010-08-25 (Estimated); Results first posted 2017-01-06 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Chronic Lymphocytic Leukemia (CLL)
Keywords: CLL; TRU-016; chronic lymphocytic leukemia; relapsed CLL; bendamustine
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — TRU 016; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase 1: 15 mg/kg TRU-016 + Bendamustine (Experimental): TRU-016 (15 mg/kg) and bendamustine (70 mg/m2), n = 6 patients
  Interventions: Drug: 15 mg/kg TRU-016 and bendamustine
- Phase 1: 20 mg/kg TRU-016 + Bendamustine (Experimental): TRU-016 (20 mg/kg) and bendamustine (70 mg/m2), n = 6 patients
  Interventions: Drug: 20 mg/kg TRU-016 and bendamustine
- Phase 2: TRU-016 and bendamustine (Experimental): TRU-016 (20 mg/kg) and bendamustine (70 mg/m2), n = 32 patients
  Interventions: Drug: TRU-016 and bendamustine
- Phase 2: Bendamustine (Active Comparator): Bendamustine (70 mg/m2), n = 33 patients
  Interventions: Drug: Bendamustine

INTERVENTIONS:
Drug: TRU-016 and bendamustine — TRU-016 at 20 mg/kg, weekly by IV infusion x 2 cycles, then every 14 days x 4 cycles PLUS bendamustine (70 mg/m2 by IV infusion on Days 1 and 2 of every 28-day cycle, for 6 cycles
  Arms: Phase 2: TRU-016 and bendamustine
Drug: Bendamustine — Bendamustine at 70 mg/m2 by IV infusion on Days 1 and 2 of every 28-day cycle, for 6 cycles
  Arms: Phase 2: Bendamustine
Drug: 15 mg/kg TRU-016 and bendamustine — TRU-016 at 15 mg/kg, weekly by IV infusion x 2 cycles, then every 14 days x 4 cycles PLUS bendamustine (70 mg/m2 by IV infusion on Days 1 and 2 of every 28-day cycle, for 6 cycles
  Arms: Phase 1: 15 mg/kg TRU-016 + Bendamustine
Drug: 20 mg/kg TRU-016 and bendamustine — TRU-016 at 20 mg/kg, weekly by IV infusion x 2 cycles, then every 14 days x 4 cycles PLUS bendamustine (70 mg/m2 by IV infusion on Days 1 and 2 of every 28-day cycle, for 6 cycles
  Arms: Phase 1: 20 mg/kg TRU-016 + Bendamustine

SUMMARY:
The objective of the first part of the study is to determine a safe dose of TRU-016 that can be used in combination with bendamustine in patients with relapsed CLL. The objectives of the second part of the study are to compare the safety and efficacy of TRU-016 in combination with bendamustine to bendamustine alone in patients with relapsed CLL.

DETAILED DESCRIPTION:
This study consisted of two parts. The initial dose escalation stage was a Phase 1b study evaluating the safety and tolerability of two doses of TRU-016 administered in combination with bendamustine to patients with relapsed chronic lymphocytic leukemia (CLL). In the randomized Phase 2 stage of the study, the efficacy and safety of the selected dose of 20 mg/kg TRU-016 combined with bendamustine was compared to bendamustine alone. The pharmacokinetics and pharmacodynamics of TRU-016 and the development of antibodies to TRU-016 were evaluated in both phases of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsed CLL with 1 to 3 prior treatments
* Demonstrated active disease requiring treatment
* No prior bendamustine treatment
* Not refractory to fludarabine or other purines, either as a single agent or in combination
* Age >/=18 years; male or female
* Eastern Cooperative Oncology Group (ECOG) performance status of </= 2
* Creatinine clearance > 40 mL/min
* Absolute neutrophil count (ANC) >/= 1,200/mm3
* Platelets >/= 75,000/mm3
* Lymphocytes >/= 5,000/mm3 in Phase 1b

Exclusion Criteria:

* Treatment with rituximab or other B-cell depleting agent within 30 days or alemtuzumab within 12 weeks
* Previous anticancer therapy within 30 days
* Refractory to prior fludarabine or other purine analog therapy either as a single agent or in combination
* Receipt of prior bendamustine or TRU-016
* Receipt of an investigational therapy or major surgery within 30 days
* Previous or concurrent additional malignancy (some exceptions apply)
* Any significant concurrent medical diseases or conditions
* Positive serology for HIV or hepatitis C, hepatitis B surface antigen positive or hepatitis B core antibody positive.
* Pregnant or breast feeding
* Drug or alcohol abuse
* Allergic to mannitol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2010-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Stromatt, MD, Study Director — Emergent Product Development Seattle LLC
Locations (25):
- United States (9):
  - For additional information regarding sites for this trial call (919) 465-4648, Denver, Colorado
  - For additional information regarding sites for this trial call (919) 465-4648, Augusta, Georgia
  - For additional information regarding sites for this trial call (919) 465-4648, Chicago, Illinois
  - For additional information regarding sites for this trial call (919) 465-4648, Hackensack, New Jersey
  - For additional information regarding sites for this trial call (919) 465-4648, Syracuse, New York
  - For additional information regarding sites for this trial call (919) 465-4648, Durham, North Carolina
  - For additional information regarding sites for this trial call (919) 465-4648, Cleveland, Ohio
  - For additional information regarding sites for this trial call (919) 465-4648, Columbus, Ohio
  - For additional information regarding sites for this trial call (919) 465-4648, Seattle, Washington
- For additional information regarding sites for this trial call (919) 465-4648, Vienna, Austria
- Germany (8):
  - For additional information regarding sites for this trial call (919) 465-4648, Bremen
  - For additional information regarding sites for this trial call (919) 465-4648, Cologne
  - For additional information regarding sites for this trial call (919) 465-4648, Frankfurt
  - For additional information regarding sites for this trial call (919) 465-4648, Göttingen
  - For additional information regarding sites for this trial call (919) 465-4648, Kiel
  - For additional information regarding sites for this trial call (919) 465-4648, Mainz
  - For additional information regarding sites for this trial call (919) 465-4648, Mutlangen
  - For additional information regarding sites for this trial call (919) 465-4648, Regensburg
- Poland (5):
  - For additional information regarding sites for this trial call (919) 465-4648, Bialystok
  - For additional information regarding sites for this trial call (919) 465-4648, Gdansk
  - For additional information regarding sites for this trial call (919) 465-4648, Lodz
  - For additional information regarding sites for this trial call (919) 465-4648, Poznan
  - For additional information regarding sites for this trial call (919) 465-4648, Warsaw
- Spain (2):
  - For additional information regarding sites for this trial call (919) 465-4648, Madrid
  - For additional information regarding sites for this trial call (919) 465-4648, Navarre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robak T, Hellmann A, Kloczko J, Loscertales J, Lech-Maranda E, Pagel JM, Mato A, Byrd JC, Awan FT, Hebart H, Garcia-Marco JA, Hill BT, Hallek M, Eisenfeld AJ, Stromatt SC, Jaeger U. Randomized phase 2 study of otlertuzumab and bendamustine versus bendamustine in patients with relapsed chronic lymphocytic leukaemia. Br J Haematol. 2017 Feb;176(4):618-628. doi: 10.1111/bjh.14464. Epub 2016 Dec 15. PMID 27977057
- See also: Otlertuzumab and Bendamustine in Relapsed CLL — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5324531/

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 15 mg/kg: TRU-016 (15 mg/kg), weekly by IV infusion x 2 cycles, then every 14 days x 4 cycles and bendamustine (70 mg/m2 by IV infusion on Days 1 and 2 of every 28-day cycle, for 6 cycles
- Phase 1 20 mg/kg: TRU-016 (20 mg/kg), weekly by IV infusion x 2 cycles, then every 14 days x 4 cycles and bendamustine (70 mg/m2 by IV infusion on Days 1 and 2 of every 28-day cycle, for 6 cycles
- Phase 2 TRU-016 and Bendamustine: Patients in the combination arm received otlertuzumab (20 mg/kg) weekly by IV infusion for two 28-day cycles then every 14 days for four 28-day cycles. In both arms, bendamustine (70 mg/m2) was administered IV on Days 1 and 2 of each cycle for up to six 28-day cycles.
- Phase 2 Bendamustine: Patients in the bendamustine arm received bendamustine (70 mg/m2) administered IV on Days 1 and 2 of each cycle for up to six 28-day cycles.
Period: Overall Study
Arm/Group | Phase 1 15 mg/kg | Phase 1 20 mg/kg | Phase 2 TRU-016 and Bendamustine | Phase 2 Bendamustine
Started | 6 | 6 | 33 (33 patients enrolled, 32 patients treated. One patient had bladder cancer and was not treated.) | 34 (34 patients enrolled, 33 patients treated. One patient withdrew consent and was not treated.)
Completed | 6 | 6 | 32 | 33
Not Completed | 0 | 0 | 1 | 1
Not completed — bladder cancer | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: patients with relapsed chronic lymphocytic leukemia
Groups:
- Phase 1: 15 mg/kg TRU-016: TRU-016 (15 mg/kg) and bendamustine (70 mg/m2)
  TRU-016 and bendamustine: TRU-016 (20 mg/kg) weekly by IV infusion x 2 cycles, then every 14 days x 4 cycles PLUS bendamustine (70 mg/m2 by IV infusion on Days 1 and 2 of every 28-day cycle, for 6 cycles
- Phase 1: 20 mg/kg TRU-016; Phase 2: TRU-016 and Bendamustine: TRU-016 (20 mg/kg) and bendamustine (70 mg/m2)
  TRU-016 and bendamustine: TRU-016 (20 mg/kg) weekly by IV infusion x 2 cycles, then every 14 days x 4 cycles PLUS bendamustine (70 mg/m2 by IV infusion on Days 1 and 2 of every 28-day cycle, for 6 cycles
- Phase 2: Bendamustine: Bendamustine alone (70 mg/m2)
  Bendamustine: 70 mg/m2 by IV infusion on Days 1 and 2 of every 28-day cycle, for 6 cycles
- Total: Total of all reporting groups
Arm/Group | Phase 1: 15 mg/kg TRU-016 | Phase 1: 20 mg/kg TRU-016 | Phase 2: TRU-016 and Bendamustine | Phase 2: Bendamustine | Total
Number analyzed (Participants) | 6 | 6 | 32 | 33 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 16 | 21 | 41
  >=65 years | 5 | 3 | 16 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (5.8) | 67.7 (8.9) | 64.1 (9.4) | 62.2 (8.1) | 62.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 12 | 8 | 24
  Male | 4 | 4 | 20 | 25 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 32 | 33 | 77
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 1 | 5
  White | 5 | 5 | 30 | 32 | 72
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Response Per International Workshop on Chronic Lymphocytic Leukemia (IWCLL) Criteria
Description: Patients had full clinical response assessment monthly during treatment, at the end of treatment (EOT) visit, 30 and 60 days after the EOT visit, and subsequently every 3 months until the earliest of progression of CLL, death, initiation of new therapy, withdrawal from the study, or completion of 18 months of follow-up evaluations. Clinical response assessment included physical examination with measurement of spleen, liver, and lymph nodes, disease-related symptoms, and laboratory measurements, specifically complete blood count (CBC) with differential.
Time Frame: 1 and 2 months after end of treatment, then every 3 months until disease progression, death, initiation of new therapy, study withdrawal, or 2 years
Population: Treated patients
Measure: Number; unit: percentage of patients
Groups:
- Phase 1 15 mg/kg TRU-016: 15 mg/kg TRU-016 + 70 mg/m2 bendamustine (n=6) dose group
- Phase 1 20 mg/kg TRU-016: 20 mg/kg TRU-016 + 70 mg/m2 bendamustine (n=6) dose group
- TRU-016 and Bendamustine: TRU-016 (n = 32 patients), 20 mg/kg and bendamustine (70 mg/m2)
  TRU-016 and bendamustine: TRU-016 (n = 33 patients), 20 mg/kg, weekly by IV infusion x 2 cycles, then every 14 days x 4 cycles PLUS bendamustine (70 mg/m2 by IV infusion on Days 1 and 2 of every 28-day cycle, for 6 cycles
- Bendamustine: Bendamustine alone (n = 33 patients) (70 mg/m2)
  Bendamustine: 70 mg/m2 by IV infusion on Days 1 and 2 of every 28-day cycle, for 6 cycles
Arm/Group | Phase 1 15 mg/kg TRU-016 | Phase 1 20 mg/kg TRU-016 | TRU-016 and Bendamustine | Bendamustine
Number analyzed (Participants) | 6 | 6 | 32 | 33
percentage of patients | 66.7 | 83.3 | 68.8 | 39.4

2. Secondary Outcome: Response Per NCI Criteria
Description: Overall response rate per National Cancer Institute (NCI) Working group criteria.
Time Frame: as for outcome 1
Population: Safety data for all patients who received any study drug and efficacy data for randomized patients who received some study treatment and have some post baseline data are presented here.
Measure: Number; unit: percentage of patients
Groups:
- Phase 2: TRU-016 and Bendamustine: TRU-016 (n = 32 patients), 20 mg/kg and bendamustine (70 mg/m2)
  TRU-016 and bendamustine: TRU-016 (n = 33 patients), 20 mg/kg, weekly by IV infusion x 2 cycles, then every 14 days x 4 cycles PLUS bendamustine (70 mg/m2 by IV infusion on Days 1 and 2 of every 28-day cycle, for 6 cycles
- Phase 2: Bendamustine: Bendamustine alone (n = 33 patients) (70 mg/m2)
  Bendamustine: 70 mg/m2 by IV infusion on Days 1 and 2 of every 28-day cycle, for 6 cycles
- Phase 1: 15 mg/kg TRU-016 +Beendamustine: TRU-016 and bendamustine: TRU-016 (n = 6 patients), 15 mg/kg, weekly by IV infusion x 2 cycles, then every 14 days x 4 cycles PLUS bendamustine (70 mg/m2 by IV infusion on Days 1 and 2 of every 28-day cycle, for 6 cycles
- Phase 1: 20 mg/kg TRU-016 +Bendamustine: TRU-016 and bendamustine: TRU-016 (n = 6 patients), 20 mg/kg, weekly by IV infusion x 2 cycles, then every 14 days x 4 cycles PLUS bendamustine (70 mg/m2 by IV infusion on Days 1 and 2 of every 28-day cycle, for 6 cycles
Arm/Group | Phase 2: TRU-016 and Bendamustine | Phase 2: Bendamustine | Phase 1: 15 mg/kg TRU-016 +Beendamustine | Phase 1: 20 mg/kg TRU-016 +Bendamustine
Number analyzed (Participants) | 32 | 33 | 6 | 6
percentage of patients | 81.3 | 66.7 | 66.7 | 100

ADVERSE EVENTS:
Time Frame: Adverse event information was collected during the clinical trial from the time consent was given through 30 days post last drug infusion.
Groups:
- Phase 1: 15 mg/kg: TRU-016 (15 mg/kg), weekly by IV infusion x 2 cycles, then every 14 days x 4 cycles PLUS bendamustine (70 mg/m2 by IV infusion on Days 1 and 2 of every 28-day cycle, for 6 cycles
- Phase 1: 20 mg/kg: TRU-016 (20 mg/kg), weekly by IV infusion x 2 cycles, then every 14 days x 4 cycles PLUS bendamustine (70 mg/m2 by IV infusion on Days 1 and 2 of every 28-day cycle, for 6 cycles
- Phase 2:Bendamustine: Bendamustine alone (70 mg/m2)
  Bendamustine: 70 mg/m2 by IV infusion on Days 1 and 2 of every 28-day cycle, for 6 cycles
Arm/Group | Phase 1: 15 mg/kg | Phase 1: 20 mg/kg | Phase 2: TRU-016 and Bendamustine | Phase 2:Bendamustine
Serious Adverse Events (participants affected / at risk) | 3/6 | 1/6 | 10/32 | 15/33
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 24/32 | 25/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: 15 mg/kg (N=6) | Phase 1: 20 mg/kg (N=6) | Phase 2: TRU-016 and Bendamustine (N=32) | Phase 2:Bendamustine (N=33)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Aplasia pure red cell (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 3 | 3
Chills (General disorders) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 3 | 4
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 3
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Thrombophlebitis septic (Infections and infestations) | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: 15 mg/kg (N=6) | Phase 1: 20 mg/kg (N=6) | Phase 2: TRU-016 and Bendamustine (N=32) | Phase 2:Bendamustine (N=33)
Neutropenia (Blood and lymphatic system disorders) | 5 | 4 | 19 | 13
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 10 | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 11 | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2
Nausea (Gastrointestinal disorders) | 5 | 5 | 6 | 10
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 5 | 7
Constipation (Gastrointestinal disorders) | 3 | 0 | 2 | 8
Vomiting (Gastrointestinal disorders) | 1 | 1 | 4 | 5
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Pyrexia (General disorders) | 1 | 3 | 11 | 4
Fatigue (General disorders) | 1 | 2 | 5 | 5
Chills (General disorders) | 1 | 2 | 4 | 2
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 2 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 4 | 7
Pneumonia (Infections and infestations) | 1 | 0 | 3 | 5
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 5 | 3
Nasopharyngitis (Infections and infestations) | 0 | 1 | 3 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 3 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 1
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 2
Weight decreased (Investigations) | 1 | 0 | 2 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 3
Hypokalaemia (Investigations) | 3 | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Headache (Nervous system disorders) | 2 | 2 | 2 | 5
Dizziness (Nervous system disorders) | 2 | 2 | 1 | 4
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 4 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 5 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 2
Hypotension (Vascular disorders) | 1 | 1 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No